CLINICAL TRIAL: NCT04406038
Title: A Population-Based Seroprevalence of SARS-CoV-2-Specific Antibodies Among Adults in Saint Petersburg, Russia: Longitudinal Cohort Study
Brief Title: Study of the Spread of COVID-19 in Saint Petersburg, Russia
Status: Completed | Type: Observational
Sponsor: European University at St. Petersburg (Other)
Responsible Party: Sponsor
Other Study IDs: CDRU-001
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: COVID19
Keywords: seroprevalence; covid-19; sars-cov-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Healthy adults randomly sampled from the population of Saint Petersburg

SUMMARY:
Seroprevalence study of COVID-19 in Saint Petersburg, Russia is a regional longitudinal cohort study aiming to evaluate the spread dynamics of the COVID-19 disease in the population of Saint Petersburg. Clinically asymptomatic adults are sampled from the population using random digit dialing and tested for the presence of SARS-CoV-2-specific antibodies in the blood serum. Data collection and serial sampling of the same individuals spans four weeks and is conducted every two weeks in order to understand both the spread of the virus in the population.

DETAILED DESCRIPTION:
At least 1 000 individuals, 18 years old and older, are randomly sampled using random digit dialing from the population of Saint Petersburg, Russia. Random sampling is performed by a survey company on the list of mobile phone numbers with designated geography prefixes of St. Petersburg. The baseline questionnaire for computer-assisted telephone interview includes travel history, medical history, and socio-economic status of the respondents. Sampled individuals are then invited to the clinic for blood sampling, their refusal to participate is recorded. Collected blood samples are used for SARS-CoV-2-specific antibodies testing. Data and sample collection spans four weeks and is conducted every two weeks. Participants complete additional questionnaires in the clinic providing information on medical history, history of allergies, chronic disease, smoking, and medication taken regularly. Contact tracing data and environmental conditions of the household are reсorded.

ELIGIBILITY:
Inclusion Criteria:

* Individuals sampled from the population of Saint Petersburg, Russia using random digit dialling.
* Subjects aged 18 and older of both genders.
* Asymptomatic at the time of blood draw.
* Written informed consent for a blood draw, SARS-COV-2 antibody test, and data collection.

Exclusion Criteria:

* Presence of fever or cough or respiratory distress at the time of blood test not attributable to other known chronic disease.
* Age under 18.
* Any health condition that may be a contraindication towards blood sampling in out-patient clinic.
* Residence in Kolpinskiy, Kurortniy, Krasnoselsky, Kronshtadtskiy, Petrodvorcoviy, Pushkinskiy districts of St. Petersburg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Representative sample of the population of Saint Petersburg, Russia
Sampling Method: Non-Probability Sample
Enrollment: 1038 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of the SARS-COV-2 infection in Saint Petersburg, Russia | Measured with two-week (14 days) intervals
  Measured by SARS-CoV-2-specific antibodies serial testing and corrected for volunteer bias and test characteristics.

SECONDARY OUTCOMES:
Prevalence odds ratios | Measured with two-week (14 days) intervals
  Comparison of prevalence by age, sex and socioeconomic strata.
Immune response dynamics | Measured with two-week (14 days) intervals
  Seropositivity, seroreversion and seroconversion.

CONTACTS AND LOCATIONS:
Overall Officials: Lubov Barabanova, MD, Principal Investigator — Clinic "Scandinavia"
Locations (1):
- Clinic "Scandinavia", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual phone survey data, anonymized paper-based survey data, test results, and analytic code are available in a designated repository (see the URL below).
Supporting Information: Analytic Code
Time Frame: Currently available and for indefinite period
Access Criteria: Creative Commons License Attribution 4.0 International (CC BY 4.0)
URL: https://github.com/eusporg/spb_covid_study20

REFERENCES:
- [Background] Barchuk A, Shirokov D, Sergeeva M, Tursun Zade R, Dudkina O, Tychkova V, Barabanova L, Skougarevskiy D, Danilenko D. Evaluation of the performance of SARS--CoV--2 antibody assays for a longitudinal population-based study of COVID--19 spread in St. Petersburg, Russia. J Med Virol. 2021 Oct;93(10):5846-5852. doi: 10.1002/jmv.27126. Epub 2021 Jun 12. PMID 34081328
- [Background] Barchuk A, Bulina A, Cherkashin M, Berezina N, Rakova T, Kuplevatskaya D, Stanevich O, Skougarevskiy D, Okhotin A. COVID-19 vaccines effectiveness against symptomatic SARS-CoV-2 during Delta variant surge: a preliminary assessment from a case-control study in St. Petersburg, Russia. BMC Public Health. 2022 Sep 22;22(1):1803. doi: 10.1186/s12889-022-14202-9. PMID 36138385
- [Background] Barchuk A, Cherkashin M, Bulina A, Berezina N, Rakova T, Kuplevatskaya D, Stanevich O, Skougarevskiy D, Okhotin A. Vaccine effectiveness against referral to hospital after SARS-CoV-2 infection in St. Petersburg, Russia, during the Delta variant surge: a test-negative case-control study. BMC Med. 2022 Sep 20;20(1):312. doi: 10.1186/s12916-022-02509-8. PMID 36123681
- [Background] Barchuk A, Bulina A, Cherkashin M, Berezina N, Rakova T, Kuplevatskaya D, Skougarevskiy D, Okhotin A. Gam-COVID-Vac, EpiVacCorona, and CoviVac effectiveness against lung injury during Delta and Omicron variant surges in St. Petersburg, Russia: a test-negative case-control study. Respir Res. 2022 Oct 10;23(1):276. doi: 10.1186/s12931-022-02206-3. PMID 36217139
- [Result] Barchuk A, Skougarevskiy D, Titaev K, Shirokov D, Raskina Y, Novkunkskaya A, Talantov P, Isaev A, Pomerantseva E, Zhikrivetskaya S, Barabanova L, Volkov V. Seroprevalence of SARS-CoV-2 antibodies in Saint Petersburg, Russia: a population-based study. Sci Rep. 2021 Jun 21;11(1):12930. doi: 10.1038/s41598-021-92206-y. PMID 34155259
- [Result] Barchuk A, Skougarevskiy D, Kouprianov A, Shirokov D, Dudkina O, Tursun-Zade R, Sergeeva M, Tychkova V, Komissarov A, Zheltukhina A, Lioznov D, Isaev A, Pomerantseva E, Zhikrivetskaya S, Sofronova Y, Blagodatskikh K, Titaev K, Barabanova L, Danilenko D. COVID-19 pandemic in Saint Petersburg, Russia: Combining population-based serological study and surveillance data. PLoS One. 2022 Jun 15;17(6):e0266945. doi: 10.1371/journal.pone.0266945. eCollection 2022. PMID 35704649
- Available data/document: Individual Participant Data Set: ID — http://github.com/eusporg/spb_covid_study20 — Please consult with the README.md for the repository.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT04406038/Prot_ICF_000.pdf